CLINICAL TRIAL: NCT07019935
Title: Afterload Mismatch Predictive modLE for Transcatheter Edge-to-Edge Repair (AMPLE-TEER Study)
Brief Title: Afterload Mismatch Predictive modLE for Transcatheter Edge-to-Edge Repair (AMPLE-TEER)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Dr., Sun Yat-sen University
Other Study IDs: AMPLE-TEER study
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Mitral Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing TEER: Adult MR patients undergoing TEER during hospitalization

SUMMARY:
Mitral regurgitation (MR) is one of the most common valvular heart diseases in China, causing heart failure. Patients with moderate to severe MR have a very poor clinical prognosis if no intervention is performed. When symptoms are still poorly controlled after guideline-directed medical therapy (GDMT) or when surgical intervention is not suitable, transcatheter mitral valve edge-to-edge repair (TEER) can improve the patient's quality of life and reduce the hospitalization rate and mortality rate. However, some patients develop into afterload mismatch (AM) after TEER, persistent adverse ventricular remodeling, and a high mortality rate, which limits the surgical benefits of TEER surgery in these MR patients. Therefore, how to scientifically predict AM and intervene as early as possible has become a research hotspot for optimizing the postoperative management of TEER patients. Afterload Mismatch Predictive modLE for Transcatheter Edge-to-Edge Repair (AMPLE-TEER) study is a prospective cohort study including adult patients undergoing TEER during hospitalization. We aim to evaluate whether the patients develop into AM after TEER, evaluate the prognostic risk factors of AM and construct a prognostic clinical model to guide clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transcatheter mitral valve edge-to-edge repair (TEER) during hospitalization.
* Aged over 18 yrs.

Exclusion Criteria:

* Patients unable to provide written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing transcatheter mitral valve edge-to-edge repair (TEER) during hospitalization were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Afterload mismatch | Through study completion, an average of 5 years
  The increase in the patient's left ventricular end-diastolic volume index (LVEDVi) after transcatheter mitral valve edge-to-edge repair (TEER) was 10% or more compared with before (dLVEDVi ≥10%).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No